CLINICAL TRIAL: NCT06915506
Title: The Effect of Shenfu Injection on Carotid Artery Elasticity in Septic Shock Patients: A Prospective Observational Pilot Study
Brief Title: Shenfu Injection Modulates Carotid Elasticity in Septic Shock
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Wuhu City Second People's Hospital (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202506
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock; Vascular Dysfunction; Arterial Stiffness; Carotid Artery Elasticity Alterations; Sepsis
Keywords: Septic shock; Shenfu Injection; Carotid artery elasticity; Ultrasound speckle tracking; Vascular dysfunction; Arterial stiffness; Strain imaging; Traditional Chinese Medicine (TCM); Circumferential strain (CS); Sepsis-associated vascular injury
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Shen-Fu

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shenfu Injection Group (Experimental): Treatment will be conducted in accordance with international and Chinese guidelines for sepsis. Following completion of fluid resuscitation and confirmation of hemodynamic stability (maintained for ≥1 hour with vasoactive agents), Shenfu Injection will be administered at a dose of 60 mL via continuous infusion over 3 hours using a syringe pump. Carotid artery circumferential strain will be quantitatively assessed using ultrasound Speckle Tracking Imaging (STI) at the following five time points to evaluate carotid artery elasticity:
  T0: Pre-administration baseline T1: 1 hour post-administration initiation T2: 2 hours post-administration initiation T3: 3 hours post-administration initiation (end of infusion) T4: 1 hour post-infusion completion
  Interventions: Drug: Shenfu Injection
- Control Group (No Intervention): Patients in this group will receive standard sepsis management strictly adhering to international and Chinese guidelines. Following completion of fluid resuscitation and confirmation of hemodynamic stability (defined as ≥1 hour of stable vasoactive agent requirements without dose escalation), carotid artery circumferential strain will be serially assessed using ultrasound speckle tracking imaging (STI) to evaluate vascular elasticity. Measurements will be performed at five predefined time points aligned with the intervention group's protocol:
  T0: Baseline (immediately post-stabilization) T1: 1 hour post-T0 T2: 2 hours post-T0 T3: 3 hours post-T0 T4: 4 hours post-T0

INTERVENTIONS:
Drug: Shenfu Injection — This intervention combines traditional Chinese medicine (TCM) with modern critical care practices to distinguish it from conventional sepsis therapies. Key unique features include:
  TCM-Based Intervention:
  Shenfu Injection: A standardized herbal extract derived from Panax ginseng and Aconitum carmichaelii , prepared under Chinese Pharmacopoeia guidelines.
  Mechanism: Targets mitochondrial dysfunction and endothelial glycocalyx repair, with preclinical evidence of anti-inflammatory, anti-apoptotic, and vasoregulatory effects.
  Precision Delivery Protocol:
  Dosage: 60 mL (1 mL/kg for patients <60 kg) administered via syringe pump-controlled continuous infusion over 3 hours, ensuring stable plasma concentrations.
  Timing: Initiated only after hemodynamic stabilization (≥1 hour of stable vasopressor requirements post-fluid resuscitation), aligning with the "golden window" for vascular repair in sepsis.
  Arms: Shenfu Injection Group

SUMMARY:
What is this study about? We are studying whether Shenfu Injection (a traditional Chinese herbal medicine) can help improve blood vessel health in patients with septic shock-a severe complication of infections that can damage blood vessels and organs. Specifically, we want to see if this treatment makes the carotid artery (a major neck blood vessel) more flexible and resilient, which may support recovery.

Who can join? Adults (18 years or older) diagnosed with septic shock by their doctors. Patients whose doctors plan to use Shenfu Injection as part of their treatment. Patients who agree to participate and sign a consent form. Who cannot join? Patients with severe heart conditions, advanced organ failure, or major neck artery disease.

Pregnant or breastfeeding women. Those unable to complete the study procedures. What will happen during the study?

Safe and Pain-Free Tests:

Ultrasound scans: A non-invasive imaging method will be used to measure the flexibility and blood flow of your neck artery.

Advanced imaging technology: A special ultrasound technique (called speckle tracking) will take detailed pictures of your artery's movement during heartbeat cycles.

Timing of Tests:

Scans will be done before receiving Shenfu Injection and 1, 2, 3 hours after the injection, plus 1 hour after treatment ends.

Other Data Collection:

Blood tests to check inflammation and organ function. Recording your health status (e.g., blood pressure, heart rate) and recovery progress (e.g., time in the Intensive Care Unit (ICU), survival rates).

What are the benefits and risks? Benefits: This study may help doctors better understand how Shenfu Injection works and improve future care for septic shock patients.

Risks: The ultrasound scans are routine, safe, and painless. There is no extra risk beyond standard hospital care.

Your Rights and Safety Voluntary Participation: You can withdraw at any time without affecting your treatment.

Ethical Approval: This study is reviewed and approved by the hospital's ethics committee.

Privacy: Your personal information and test results will be kept confidential.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Diagnosis of sepsis or septic shock in the acute phase, as defined by the -Sepsis-3 criteria (confirmed infection with Sequential Organ Failure Assessment [SOFA] score ≥ 2 points above baseline).
* Voluntary participation with written informed consent provided by the patient or legally authorized representative.

Exclusion Criteria

* Severe carotid atherosclerosis (e.g., carotid Intima-Media Thickness (IMT)>1.2 mm or confirmed plaque formation) diagnosed by prior imaging.
* Significant cardiovascular comorbidities that may confound hemodynamic assessments, including:
* Severe cardiomyopathy (e.g., ejection fraction <30%).
* Uncontrolled arrhythmias (e.g., ventricular tachycardia, atrial fibrillation with rapid ventricular response).
* Congenital heart disease with hemodynamic instability.
* Active hepatic or renal insufficiency (e.g., Child-Pugh class C, dialysis dependence) or advanced systemic diseases (e.g., metastatic malignancy, terminal illness).
* Poor ultrasound image quality precluding reliable speckle tracking analysis (e.g., inadequate acoustic window, motion artifacts).
* Pregnancy or lactation (due to potential hormonal influences on vascular physiology).
* Withdrawal from the study or inability to complete follow-up assessments (e.g., non-compliance, transfer to another facility).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Carotid Artery Circumferential Strain (CS) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Peak deformation of the carotid artery wall during the cardiac cycle, measured via ultrasound speckle tracking imaging (STI).Derived from strain rate analysis using dedicated vascular ultrasound software.
Carotid Artery Elasticity (Beta (β)2 Stiffness Index) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Description: Composite metric integrating blood pressure and circumferential strain to quantify vascular stiffness.
  Calculation: β 2= ln(Systolic Blood Pressure/Diastolic Blood Pressure)/CS Data Sources: Blood pressure (non-invasive monitoring) + STI-derived CS.

SECONDARY OUTCOMES:
Carotid Artery Elasticity (β1 Stiffness Index) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Calculation：β 1 = ln(Systolic Blood Pressure/Diastolic Blood Pressure)/(Ds-Dd)×Dd
Carotid Artery Systolic Diameter (Ds) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Maximum diameter during systole (millimeters, mm)
Carotid Artery Diastolic Diameter (Dd) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Minimum diameter during diastole (millimeters, mm)
Carotid Artery Peak Systolic Velocity (PSV) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Parameter: Maximum flow velocity during systole by Doppler Ultrasound Unit: cm/s Measurement**: Pulsed-wave Doppler spectral analysis
Carotid Artery End-Diastolic Velocity (EDV) | T0: Baseline (pre-treatment); T1: 1 hour after initiation of Shenfu Injection/control protocol ;T2: 2 hours after initiation; T3: 3 hours after initiation (end of infusion) ;T4: 1 hour post-infusion completion
  Parameter: Minimum flow velocity at end-diastole by Doppler Ultrasound Unit: cm/s Measurement**: Pulsed-wave Doppler spectral analysis
ICU Length of Stay | up to 28 days
  Days from enrollment to ICU discharge.
28-Day All-Cause Mortality | Day 28 post-enrollment
  Survival status at 28 days post-enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital of Wannan Medical College), Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes